CLINICAL TRIAL: NCT00119938
Title: D-STAR (Diabetes-System To Access Records): An Online Patient Portal to Improve and Sustain Diabetes Self-Care
Brief Title: An Online System to Improve Diabetes Self-Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 51758
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2007-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Disease management; Patient access to records; Medical records systems, computerized; Questionnaires; Physician-patient relations; Medical records
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Access to online patient portal

SUMMARY:
The purpose of this study is to see if an online program for patients with diabetes helps patients improve their self-care (how they take their medications, what they eat, how much they exercise, and whether they smoke).

DETAILED DESCRIPTION:
Patient portals are online programs that can provide a number of functions for patients, among them:

* Ability to request appointments, referrals, and medication refills;
* Ability to send secure electronic messages to medical staff, and to receive replies;
* Access to the medical record;
* Disease management

We are comparing two patient portals with different sets of features to determine if personalized information and guidance can improve self-care and measures of diabetes-related health. Self-care measures will be assessed using standardized questionnaires at baseline, 3, and 6 months. Chart review will be used to assess measures of diabetes-related health.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 diabetes mellitus
* Has access to Internet
* Has e-mail address
* Established patient at one of four participating practices at University of Colorado Hospital

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2004-09; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Composite measure of diabetes self-care activities, developed from the Summary of Diabetes Self-Care Measure | Surveys at baseline, 3 months, and 6 months

SECONDARY OUTCOMES:
Qualitative assessment of the program by patients and medical staff | Interviews after 9 months of deployment
Biological markers of diabetes care (hemoglobin A1c, blood pressure, LDL cholesterol) | Incidentally obtained over 9 months of care

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Ross, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- See also: Website for Health e-Technologies Initiative, a national program office of the Robert Wood Johnson Foundation — http://www.hetinitiative.org
- See also: Website for University of Colorado Hospital, the site of the study — http://www.uch.edu